CLINICAL TRIAL: NCT04230499
Title: Phase IIA Trial of Encapsulated Rapamycin (eRapa) to Prevent Progression in Familial Adenomatous Polyposis Patients Under Active Surveillance
Brief Title: Trial of ERapa to Prevent Progression in Familial Adenomatous Polyposis Patients Under Active Surveillance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rapamycin Holdings Inc. (Industry)
Collaborators: Cancer Insight, LLC (Industry); Biodexa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EMT-FAP-001
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-10

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Intervention Model Description: Patients will receive one of three doses in a dose-escalating fashion. Cohort 1 will receive 0.5mg every other day, Cohort 2 will receive 0.5mg daily with 7 days on therapy followed by 7 days off therapy, and Cohort 3 will receive 0.5 mg daily. Patients will serve as their own control; no placebo will be given.
  Additionally, a subset of participants will be included in a randomized, balanced, single-schedule, two-treatment period (fed versus fasted) crossover study.
  Participants will receive eRapa under fed or fasted conditions in the first period, and then crossover to the other treatment (fed to fasted and vice versa) following a 2 week washout. Under this design, participants serve as their own control and will allow the assessment of the effect of food on the anticipated R2PD of eRapa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will receive 0.5mg of eRapa every other day.
  Interventions: Drug: Encapsulated Rapamycin (eRapa)
- Cohort 2 (Experimental): Cohort 2 will receive 0.5mg of eRapa daily with 7 days on therapy, followed by 7 days off therapy.
  Interventions: Drug: Encapsulated Rapamycin (eRapa)
- Cohort 3 (Experimental): Cohort 3 will receive 0.5 mg of eRapa daily.
  Interventions: Drug: Encapsulated Rapamycin (eRapa)
- Food Effect (Experimental): Upon identification of the RP2D, after a 2 week washout (14 days), subjects will be randomized into a fed and fasted (2 weeks - 14 days) two period cross over, with an intervening 2 week washout (14 days) for a total of 2 months (8 weeks).
  Interventions: Drug: Encapsulated Rapamycin (eRapa)

INTERVENTIONS:
Drug: Encapsulated Rapamycin (eRapa) — eRapa is encapsulated rapamycin. The rapamycin is encapsulated in order to deliver the rapamycin at a consistent and lower dosage. eRapa is a capsule, and is administered orally.
  Other Names: eRapa; Encapsulated sirolimus

SUMMARY:
Patients with Familial Adenomatous Polyposis (FAP) who are undergoing endoscopic surveillance will be given Encapsulated Rapamycin (eRapa) at one of three escalating doses/schedules for 12 months with the aim of reducing polyp burden.

DETAILED DESCRIPTION:
Patients with FAP who are undergoing endoscopic surveillance will be given eRapa at one of three escalating doses/ schedules (0.5mg every other day, 0.5mg daily every other week, or 0.5mg daily) for 12 months with the aim of reducing polyp burden. Patients will serve as their own controls. Patients will be assessed with surveillance endoscopy at baseline, 6 months, and 12 months for change in polyp burden. Correlation between immune markers and clinical outcomes will be explored.

This is a Phase IIa trial which will enroll at approximately 6-8 sites within the United States that have specialty expertise in FAP treatment and surveillance. The trial is anticipated to last approximately 24 months for treatment and follow up.

The trial will enroll 30 patients with the genetic or clinical diagnosis of FAP. The clinical diagnosis includes individuals with 100 or more cumulative tubular adenomas throughout the colorectum. Patients must be undergoing surveillance for known FAP and can include those with intact colons as well as those who have undergone surgical therapy. For those patients who have undergone partial or total colectomy, they must have documented residual polyps in their rectum for which they are receiving active surveillance.

Once the recommended phase 2 dose (RP2D) is identified, subjects will undergo evaluation under fed and fasted states to determine the food effect on eRapa absorption.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date an informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, age at least 18 years at the time of consent.
4. Phenotypic familial adenomatous polyposis (FAP) with disease involvement of the colorectum by either genetic or clinical diagnosis: Adenomatous polyposis coli (APC) germline mutation with or without family history, or with greater than a cumulative lifetime history of (>) 100 adenomas in large intestine and a family history of FAP, or FAP phenotype post colectomy for polyposis with a family history of FAP. Minimum number of polyps required for enrollment is 10.
5. Abilitiy to safely undergo endoscopy.
6. Ability to take oral medication and be willing to adhere to the eRapa regimen.
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 12 weeks after the end of eRapa administration.
8. A woman must agree not to breast feed or donate eggs (ova, oocytes) during the study and for a period of 12 weeks after the last administration of study drug.

Exclusion Criteria:

1. Risk-reduction surgery (colectomy or partial colectomy) within the 12 months prior to screening.
2. Use of non-steroidal anti-inflammatory drugs other than aspirin during the study. The use of 81 milligrams (mg) of aspirin a day or 650 mg of aspirin per week is allowed.
3. Treatment with other FAP-directed drug therapy (including NSAID [Non-steroidal anti-inflammatory drug] drugs), unless completes a 4 week washout period prior to enrollment.
4. Duodenum or colon/ rectum with high grade dysplasia or cancer on biopsy at screening.
5. Duodenal or colorectal polyp > 1 centimeter (cm) not excised at the screening evaluation.
6. Pregnancy or breast feeding.
7. Unable to provide consent or anticipated inability to attend appropriate follow-up visits.
8. Serum creatinine or measured/ calculated creatinine clearance (or glomerular filtration rate [GFR]) > 1.5 x ULN OR < 30mL/min for participants with creatine levels > 1.5 x institutional ULN. Bilirubin ≥ 1.5 x ULN unless conjugated bilirubin ≤ ULN; alkaline phosphatase > 5 x ULN; ALT/AST > 2 x ULN.
9. INR or PT or aPTT > 1.5 x institutional ULN unless the patient is receiving anticoagulant therapy as long as the PT or aPTT is within therapeutic range of intended use of anticoagulants.
10. Proteinuria > 1+ on urinalysis or > 1g/24h on 24h urine.
11. History of interstitial lung disease or non-infectious pneumonitis.
12. Immunosuppressed state (e.g., HIV, use of chronic steroids), active, uncontrolled infection.
13. On agents known to alter rapamycin metabolism significantly.
14. Concurrent involvement in other clinical trials specifically evaluating chemoprevention in FAP.
15. Patients with a colonic polyp burden too numerous to count.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events associated with low dose eRapa in FAP patients | All adverse events with start dates occurring any time after informed consent is obtained until 7 days (for non-serious adverse events) or 30 days (for serious adverse events) after the last day of study participation will be recorded.
  Safety and tolerability of eRapa as determined by graded toxicity assessed throughout the trial per CTCAE v5.0.
Determine the Recommended Phase 2 Dose (RP2D) | After informed consent is obtained up to 30 days after the last day of study participation.
  The Recommended Phase 2 Dose (RP2D) will be determined by examining and analyzing safety/ adverse events as reflected by Outcome 1, dose delays, dose reductions, withdrawal of treatment secondary to low-grade toxicities, and serum pharmacokinetic monitoring.
Efficacy of eRapa in delaying polyp progression in patients with FAP as measured by change in polyp burden over time. | Time for each patient is baseline to 6 months.
  Percentage change from baseline in colorectal polyp burden as measure by endoscopy at 6 months.

SECONDARY OUTCOMES:
Clinical effect of eRapa on polyp burden. | Following patients out to 12 months.
  Percentage change from baseline in colorectal polyp burden at 12 months.
Clinical effect of eRapa on International Society for Gastrointestinal Hereditary Tumors Stage. | Following patients out to 6 and 12 months.
  Change from baseline in International Society for Gastrointestinal Hereditary Tumors Stage at 6 and 12 months.
Clinical effect of eRapa on Spigelman Stage Score. | Following patients out to 6 and 12 months.
  Change from baseline in Spigelman Stage Score at 6 and 12 months in patients with polyps at baseline on EGD. The Spigelman scoring system assigns points (0, 1, 2, or 3) based on number of adenomas, size (mm), histology, and dysplasia. The scoring ranges from 0 to 12 points. A higher score is a worse outcome.
Clinical effect of eRapa on duodenal polyp number and burden. | Following patients out to 6 and 12 months.
  Percentage change from baseline in the duodenal polyp number and burden at 6 and 12 months in patients with polyps at baseline on EGD.
Determine the effect of food on eRapa absorption | 2 months
  Pharmacokinetic parameters (AUC[0-INF], Cmax) to assess the effect of food on the bioavailability of the anticipated RP2D

OTHER OUTCOMES:
Explore correlation between immune markers influenced by mTOR inhibition and clinical outcomes | Following patients out to 12 months.
  Immunologic response will be measured and will include overall assessment of T cell phenotype and function.

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, Study Director — Sponsor CMO
Locations (4):
- United States (4):
  - Michigan Medicine, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - UT Health, San Antonio, Texas

REFERENCES:
- [Derived] Stone JK, Mehta NA, Singh H, El-Matary W, Bernstein CN. Endoscopic and chemopreventive management of familial adenomatous polyposis syndrome. Fam Cancer. 2023 Oct;22(4):413-422. doi: 10.1007/s10689-023-00334-3. Epub 2023 Apr 29. PMID 37119510